CLINICAL TRIAL: NCT03899558
Title: The Role of Humidified Nasal High-flow to Reduce 30-day Hospital Re-admissions Following Severe Exacerbations of Chronic Obstructive Pulmonary Disease: a Mixed Methods Feasibility Study
Brief Title: The Role of HNHF to Improve Clinical Outcomes Following Severe AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 242147
Record Dates: First submitted 2019-03-21; First posted 2019-04-02 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Neural respiratory drive; Physiology; Respiratory muscles; COPD exacerbation; Ventilation; Nasal high-flow; High-flow nasal cannula
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): HNHF device (intervention) + usual care
  Interventions: Device: Humidified nasal high-flow device
- Control (No Intervention): Usual care alone

INTERVENTIONS:
Device: Humidified nasal high-flow device — Humidified nasal high-flow device which delivers warmed, humidified air at flow rates of up to 60 litres per minute via a nasal cannula interface. Intended delivery at 30 L/min at 37 degrees Celsius, if tolerated.
  Arms: Intervention

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common lung disease, affecting 1.2 million people in the United Kingdom (UK). COPD patients suffer with episodes of worsening breathing symptoms called acute exacerbations (AECOPD). Exacerbations occur more often as the disease progresses and are a leading cause of emergency hospitalisation. Patients recovering from exacerbations are at high risk of deteriorating, with one quarter readmitted to hospital within thirty days. COPD thus imposes immense burdens on the National Health Service and patients.

This research will investigate the effects of using humidified nasal high-flow (HNHF) during recovery from severe COPD exacerbations. HNHF delivers warmed, humidified air under flows of up to 60 litres per minute through a nasal interface. This has been shown to improve clinical outcomes, including exacerbation frequency, hospitalisations, breathlessness and quality of life amongst COPD patients with respiratory failure. It is thought to achieve this by improving secretion clearance and providing positive airways pressure which supports the breathing system.

Patients admitted to St Thomas' Hospital, London with COPD exacerbations will be recruited. Prior to discharge, participants will be randomised to receive either usual care alone or usual care plus a HNHF device, which they will be trained to use for a regular period daily. Usual care includes inhalers, steroids and may include antibiotics.

Participants will be followed up for 30-days after hospital discharge using weekly assessments, daily symptom diaries and wrist-worn watch-like devices that detect physical activity. This will enable evaluation of the clinical effects of HNHF on re-exacerbations, readmissions, breathlessness, physical activity and quality of life. Device usage will also be quantified. Participants who receive devices will be interviewed to explore their experiences. After the 30-day home follow-up period, a sub-group of participants will undergo detailed breathing tests during and after exercise to explore the effects of HNHF on the respiratory system.

ELIGIBILITY:
Inclusion Criteria:

* Emergency hospital admission with a primary diagnosis of AECOPD
* Aged 40-80 years
* ≥10 pack year smoking history
* Body mass index ≤ 35kg/m2
* Cognitively and linguistically able to follow English instructions, provide informed consent and complete the study protocol
* To be discharged home following the hospitalisation in a home environment deemed safe by the investigator to perform home assessments
* Patient lives in the catchment area served by the Integrated Respiratory Team at Guy's and St Thomas' NHS Foundation Trust

Exclusion Criteria:

* Chest radiograph excludes pneumothorax
* Requirement for acute non-invasive ventilation (NIV) during index hospitalisation or established on home positive airway pressure (PAP)
* Significant chronic respiratory failure (PaCO2 >7.0)
* Clinically significant obstructive sleep apnoea requiring treatment
* Allergies to latex, metals or local anaesthetic
* Broken or inflamed skin at the second intercostal space parasternal chest wall areas
* Psychological or social factors that would impair compliance with the study protocol
* Any major non-COPD chronic co-morbidity that may contribute significantly to risk of readmission, including (but not limited to) severe heart failure (left ventricular ejection fraction <30%), malignancy (active treatment or palliation), end stage renal failure and significant neuromuscular disease
* Planned travel away from home in the 30-day post-discharge period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Time to 30-day hospital readmission following index hospitalisation with AECOPD | 30 days following hospital discharge
  30-day readmission

SECONDARY OUTCOMES:
Recruitment rate of eligible patients | 30 days following hospital discharge
  Feasibility outcome measure: assessed by proportion of patients who fulfil eligibility criteria who consent to participate.
Adherence with completion of clinical outcome measures (symptom diary) | 30 days following hospital discharge
  Feasibility outcome measure: assessed by completion of symptom diaries. Progression criterion = participant diaries completed by >70% of participants. Assessed at 30-days following hospital discharge.
Adherence with completion of clinical outcome measures (physical activity monitor) | 30 days following hospital discharge
  Feasibility outcome measure: assessed by usage of physical activity monitors. Progression criterion = usage >70% of participants. Measured from physical activity monitor computer downloads at 30-days following hospital discharge.
Adherence with completion of clinical outcome measures (spirometry) | 30 days following hospital discharge
  Feasibility outcome measure: assessed by completion of spirometry. Progression criterion = spirometry measured at every study assessment for >70% of participants.
Participants' HNHF device usage | 30 days following hospital discharge
  Feasibility outcome measure: usage hours accessed from the device at completion of participants' study participation for those participants allocated to the intervention arm.
Acceptability of HNHF at home: semi-structured interviews | 30 days following hospital discharge
  Qualitative evaluation: Use of semi-structured interviews after 30 days post-discharge following index hospitalisation to explore barriers and facilitators to device usage in intervention arm participants.
Non-readmission AECOPD | 30 days following hospital discharge
  Clinical outcome measure: the number of acute exacerbations of COPD that do not require hospitalisation will be recorded using symptom diaries.
Breathlessness | 30 days following hospital discharge
  Clinical outcome measure: breathlessness severity will be assessed using the modified Borg scale (minimum score = 0, indicating no breathlessness, maximum score = 10 indicating maximal intensity of breathlessness).
Breathlessness | 30 days following hospital discharge
  Clinical outcome measure: breathlessness severity will be assessed using the Multidimensional Dyspnoea Profile.
Physical activity | 30 days following hospital discharge
  Clinical outcome measure: daily physical activity (measured in counts per minute) will be quantified using a wrist-worn physical activity monitor which uses a triaxial accelerometer.
Health-related quality of life: COPD Assessment Test | 30 days following hospital discharge
  Clinical outcome measure: assessed using the COPD Assessment Test.
Health-related quality of life: Clinical COPD Questionnaire | 30 days following hospital discharge
  Clinical outcome measure: assessed using the Clinical COPD Questionnaire. Scored from 0 to 60, with higher scores indicative of worse disease-specific health-related quality of life.
Inspiratory capacity | 30 days following hospital discharge
  Proof of concept study outcome: measured during the physiological sub-study involving incremental exercise using a pneumotachograph.
Breathlessness | 30 days following hospital discharge
  Proof of concept study outcome: measured during the physiological sub-study involving incremental exercise using the modified Borg scale. This zero to ten scale measures breathlessness intensity, with higher scores representing more intense breathlessness. The score will be measured before exercise, at 2 minute intervals during exercise, at exercise cessation and during exercise recovery.
Neural respiratory drive | 30 days following hospital discharge
  Proof of concept study outcome: measured during the physiological sub-study involving incremental exercise using a parasternal and diaphragm electromyography using surface and nasogastric electrodes, respectively.
Pulmonary pressures and flow | 30 days following hospital discharge
  Proof of concept study outcome: measured during the physiological sub-study involving incremental exercise using a pressure transducer connected to a nasogastric catheter and a pneumotachograph.
Time to recover from maximal breathlessness | 30 days following hospital discharge
  Proof of concept study outcome: time from maximal breathlessness at peak exercise to pre-exercise modified Borg scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Suh ES, Mandal S, Harding R, Ramsay M, Kamalanathan M, Henderson K, O'Kane K, Douiri A, Hopkinson NS, Polkey MI, Rafferty G, Murphy PB, Moxham J, Hart N. Neural respiratory drive predicts clinical deterioration and safe discharge in exacerbations of COPD. Thorax. 2015 Dec;70(12):1123-30. doi: 10.1136/thoraxjnl-2015-207188. Epub 2015 Jul 20. PMID 26194996
- [Background] Murphy PB, Kumar A, Reilly C, Jolley C, Walterspacher S, Fedele F, Hopkinson NS, Man WD, Polkey MI, Moxham J, Hart N. Neural respiratory drive as a physiological biomarker to monitor change during acute exacerbations of COPD. Thorax. 2011 Jul;66(7):602-8. doi: 10.1136/thx.2010.151332. Epub 2011 May 19. PMID 21597112